CLINICAL TRIAL: NCT05968677
Title: Pragmatic, Controlled, Single-Center, Randomized Clinical Trial to Evaluate the Effect of Supplementation With an Amino Acids and Flavonoids Containing FSMP on Chemotherapy Toxicity, Nutritional Status and Quality of Life in Breast Cancer Patients
Brief Title: Effect of an Amino Acids and Flavonoids Containing FSMP on Chemotherapy Toxicity, Nutritional Status and Quality of Life in Breast Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Flavolife Srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SELECT-BC
Record Dates: First submitted 2023-07-03; First posted 2023-08-01 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: breast cancer; flavonoids; aminoacids; nutrition
MeSH Terms: conditions — Breast Neoplasms | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FSMP (Experimental): Nutritional counseling plus one sachet of the study product (6.5 g) per day, away from meals, starting the day after the first chemotherapy cycle until three weeks after the last chemotherapy cycle (for a total of 12 weeks)
  Interventions: Dietary Supplement: FSMP; Other: Nutritional counseling
- Control (Other): Nutritional counseling
  Interventions: Other: Nutritional counseling

INTERVENTIONS:
Dietary Supplement: FSMP — Food for Special Medical Purposes specifically formulated for the dietary management of malnourished patients following therapeutic treatments such as chemo and radiotherapy
  Arms: FSMP
Other: Nutritional counseling — Participant's nutritional status will be evaluated, anthropometric data will be collected (weight, height, BMI), body composition will be evaluated (FFMI, BIVA) and a food diary will be compiled

SUMMARY:
The goal of this clinical trial is to compare the effect of a Food for Special Medical Purposes (FSMP) mainly containing amino acids and flavonoids in combination with nutritional counseling, versus nutritional counseling alone, on chemotherapy toxicity, nutritional status and quality of life in patients with breast cancer.

The main questions it aims to answer are:

* can this dietary supplementation affect the nutritional status of breast cancer patients?
* can this dietary supplementation have any beneficial effect on chemotoxicity? Participants will be asked to undergo nutritional counseling and to take the study product every day for 12 weeks.

Researchers will compare a similar group of participants only receiving the nutritional counseling to see if any difference occurs.

DETAILED DESCRIPTION:
Participants will be selected at the first oncological visit at the Outpatient Clinics or the Department of Medical Oncology of the IRCCS Policlinico San Matteo of Pavia. The doctor, evaluated the inclusion and exclusion criteria, will propose patient to participate in the study and, after obtaining informed consent, will proceed with enrollment. On the first day of chemotherapy, participants will undergo an oncological and nutritional examination, with collection of anthropometric data, assessment of body composition, assessment of quality of life through special validated questionnaires, blood sampling for blood chemistry tests and urine collection. Participants in the treated group will receive a supply of the FSMP to take home. At check-up visits, the participant's nutritional status and any adverse events will be assessed, other than adherence to treatment by delivery of empty product boxes and chemotherapy compliance. Blood chemistry tests will be repeated at 6 weeks after the first chemotherapy cycle and 3 weeks after the last chemotherapy cycle (follow-up period).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-metastatic ductal breast cancer
* Post-menopausal women
* Chemotherapy with Doxorubicin or Epirubicin, with or without Cyclophosphamide, scheduled as adjuvant or neo-adjuvant
* Written informed consent
* Independent oral feeding
* Must be able to carry out periodic visits

Exclusion Criteria:

* Artificial feeding
* Eastern Cooperative Oncology Group (ECOG) performance status >2
* Impossibility to take the foreseen measurements
* Other tumor pathologies
* Previous therapy with Doxorubicin or Epirubicin
* Ongoing treatment with molecular targeted therapies
* Previous chronic renal, hepatic or cardiac insufficiency
* History of mental disorders
* Known allergies or intolerances to any study product ingredient
* Participation in other interventional clinical trials in the past three months

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-04 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in High-Sensitivity Troponin Levels as a serological marker of chemotherapy cardiotoxicity | 0, 6, 12 weeks
  The comparison of changes from baseline will be performed using a generalized linear regression model, adjusting for the baseline value of the biomarker. The difference in averages between groups and the relative range of confidence of 90 percent will be derived from the model

SECONDARY OUTCOMES:
Mean change from baseline in weight, Body Mass Index (BMI) and Fat Free Mass Index (FFMI) | 0, 3, 6, 9, 12 weeks
  Participant's weight in kilograms and height in meters will be combined to report BMI and FFMI in kg/m^2
Mean change from baseline in Phase Angle | 0, 3, 6, 9, 12 weeks
  Participant's body composition will be evaluated through measurement of the phase angle which represents the relationship between resistance and capacitive reactance of the body and bioimpedance diagnostics
Mean change from baseline in Bioelectrical Impedance Vector Analysis (BIVA) | 0, 3, 6, 9, 12 weeks
  Participant's water and nutritional status will be evaluated
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 3, 6, 9, 12 weeks
  Proportion of participants with adverse events of any type and specifically haematological, cardiac, gastrointestinal, hepatobiliary, metabolic, psychiatric, renal and urinary types, distinguishing between grade 1-2, grade 3-4 and grade 5.
  Furthermore, the proportion of participants who discontinue chemotherapy treatment and the change in the number of participants who reduce their chemotherapy dose during the treatment
Mean change from baseline in Interleukine-6 levels | 0, 6, 12 weeks
  The comparison of changes from baseline will be performed using a generalized linear regression model, adjusting for the baseline value of the biomarker. The difference in averages between groups and the relative range of confidence of 90 percent will be derived from the model
Mean change from baseline Interleukine-1 beta levels | 0, 6, 12 weeks
  The comparison of changes from baseline will be performed using a generalized linear regression model, adjusting for the baseline value of the biomarker. The difference in averages between groups and the relative range of confidence of 90 percent will be derived from the model
Mean change from baseline in C-reactive Protein levels | 0, 6, 12 weeks
  The comparison of changes from baseline will be performed using a generalized linear regression model, adjusting for the baseline value of the biomarker. The difference in averages between groups and the relative range of confidence of 90 percent will be derived from the model
Participant's perception of her physical and mental state | 0, 12 weeks
  Comparison of the total average values resulting from the compilation of two validated oncological questionnaires, which include questions with scores from 1 to 4, where in general higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pedrazzoli, MD, Principal Investigator — Unit of Medical Oncology-IRCSS San Matteo University Hospital Foundation
Locations (1):
- IRCSS San Matteo University Hospital Foundation, Pavia, Italy